CLINICAL TRIAL: NCT06941272
Title: LIGHTBEAM-U01 Substudy 01C: A Phase 1/2 Substudy to Evaluate the Safety and Efficacy of Patritumab Deruxtecan in Pediatric Participants With Relapsed or Refractory Solid Tumors
Brief Title: A Study of Patritumab Deruxtecan in Pediatric Participants With Relapsed or Refractory Solid Tumors (MK-9999-01C/LIGHTBEAM-U01)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9999-01C; MK-9999-01C (Other: MSD); LIGHTBEAM-U01 (Other: MSD); U1111-1314-1866 (Registry Identifier: UTN); 2024-518771-66-00 (Registry Identifier: EU CT)
Record Dates: First submitted 2025-02-27; First posted 2025-04-23 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Malignant Neoplasm
MeSH Terms: conditions — Neoplasms | interventions — patritumab deruxtecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Patritumab Deruxtecan (Experimental): Participants receive patritumab deruxtecan via IV infusion on Day 1 of each 3-week cycle until discontinuation or progression.
  Interventions: Biological: Patritumab Deruxtecan

INTERVENTIONS:
Biological: Patritumab Deruxtecan — IV Infusion
  Other Names: MK-1022; HER3-DXd; U3-1402

SUMMARY:
Researchers are looking for new ways to treat children with hepatoblastoma or rhabdomyosarcoma (RMS) that has relapsed or is refractory:

* Hepatoblastoma is a common liver cancer in babies and very young children
* RMS is a cancer that starts in muscle cells, often in a child's head and neck, bladder, arms, or legs
* Relapsed means the cancer came back after treatment
* Refractory means the cancer did not respond (get smaller or go away) to treatment

The study treatment HER3-DXd (also known as MK-1022 or patritumab deruxtecan) is an antibody-drug conjugate (ADC). An ADC attaches to a protein on cancer cells and delivers treatment to destroy those cells. The goals of this study are to learn:

* About the safety of HER3-DXd in children and if they tolerate it
* What happens to HER3-DXd in children's bodies over time
* If children who receive HER3-DXd have the cancer get smaller or go away

DETAILED DESCRIPTION:
This study will have 2 parts: a safety lead-in to demonstrate a tolerable safety profile and confirm a preliminary recommended phase 2 dose (RP2D) (Part 1) followed by an efficacy evaluation (Part 2)

ELIGIBILITY:
The main inclusion criteria include but are not limited to the following:

* Has one of the following histologically confirmed advanced or metastatic solid tumors: Rhabdomyosarcoma (RMS), or Hepatoblastoma
* Has progressed after at least 1 prior systemic treatment for RMS or hepatoblastoma and who has no satisfactory alternative treatment option (ie, is ineligible for other standard treatment regimens)
* Participants who have adverse events (AEs) due to previous anticancer therapies must have recovered to Grade ≤1 or baseline. Participants with endocrine-related AEs who are adequately treated with hormone replacement or participants who have Grade ≤2 neuropathy are eligible. Participants with Grade ≤2 alopecia are also eligible
* Hepatitis B surface antigen (HBsAg) positive participants are eligible if they have received hepatitis B virus (HBV) antiviral therapy and have undetectable HBV viral load
* Participants with a history of hepatitis C virus (HCV) infection are eligible if HCV viral load is undetectable

The main exclusion criteria include but are not limited to the following:

* Has a history of (noninfectious) interstitial lung disease (ILD)/pneumonitis that required steroids or has current ILD/pneumonitis, and/or suspected ILD/pneumonitis that cannot be ruled out by standard diagnostic assessments
* Has clinically severe respiratory compromise resulting from intercurrent pulmonary illness
* Has a history of solid organ transplant
* Has a history of allogeneic stem cell transplant
* Has clinically significant corneal disease
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis/leptomeningeal disease; participants with previously treated brain metastases may participate provided they are radiologically stable (ie, without evidence of progression) for at least 4 weeks
* Has uncontrolled or significant cardiovascular disorder
* Has a history of clinically significant congenital cardiac syndrome
* Has a history of human immunodeficiency virus (HIV) infection
* Has a known additional malignancy that is progressing or has required active treatment within the past 1 year
* Has an active infection requiring systemic therapy
* Has concurrent active hepatitis B (HBsAg positive and/or detectable HBV deoxyribonucleic acid [DNA]) and HCV defined as anti-HCV antibody (Ab) positive and detectable HCV ribonucleic acid [RNA]) infection
* Has not adequately recovered from major surgery or have ongoing surgical complications

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2025-05-26 (Actual); Primary Completion 2030-12-30 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
Part 1: Percentage of Participants Who Experience Dose-limiting Toxicities (DLTs) | Cycle 1 (up to approximately 21 days); each cycle is 21 days
  A DLT is any of a prespecified list of adverse events (AEs) that occur during Cycle 1 (up to 21 days) if attributed to the study treatment and not attributed to any other clearly identifiable cause. The percentage of participants who experience DLTs will be reported. Each cycle is 21 days.
Part 1: Percentage of Participants Who Experience an Adverse Event (AE) | Up to approximately 5 years
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The percentage of participants who experience AEs will be reported.
Part 1: Percentage of Participants Who Discontinue Study Treatment Due to an AE | Up to approximately 5 years
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The percentage of participants who discontinue study treatment due to an AE will be reported.
Part 1: Area Under the Curve (AUC) of total anti-HER3 antibody liquid chromatography-mass spectrometry (LC-MS) in plasma | At designated timepoints (up to approximately 5 years)
  Blood samples will be collected at specified intervals for the determination of AUC.
Part 1: AUC of anti-HER3 antibody-conjugated DXd (anti-HER3-ac-DXd) in plasma | At designated timepoints (up to approximately 5 years)
  Blood samples will be collected at specified intervals for the determination of AUC.
Part 1: AUC of DXd in plasma | At designated timepoints (up to approximately 5 years)
  Blood samples will be collected at specified intervals for the determination of AUC.
Part 1: Maximum Concentration (Cmax) of anti-HER3 antibody LC-MS in plasma | At designated timepoints (up to approximately 5 years)
  Blood samples will be collected at specified intervals for the determination of Cmax.
Part 1: Cmax of anti-HER3-ac-DXd in plasma | At designated timepoints (up to approximately 5 years)
  Blood samples will be collected at specified intervals for the determination of Cmax.
Part 1: Cmax of DXd in plasma | At designated timepoints (up to approximately 5 years)
  Blood samples will be collected at specified intervals for the determination of Cmax.
Part 1: Concentration Immediately Before the Next Dose is Administered (Ctrough) of anti-HER3 antibody LC-MS in plasma | At designated timepoints (up to approximately 5 years)
  Blood samples will be collected at specified intervals for the determination of Ctrough.
Part 1: Ctrough of anti-HER3-ac-DXd | At designated timepoints (up to approximately 5 years)
  Blood samples will be collected at specified intervals for the determination of Ctrough.
Part 1: Ctrough of DXd in plasma | At designated timepoints (up to approximately 5 years)
  Blood samples will be collected at specified intervals for the determination of Ctrough.
Part 1 and Part 2: Objective Response Rate (ORR) | Up to approximately 5 years
  ORR is defined as the percentage of participants with Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST 1.1). The percentage of participants who experience CR or PR as assessed by the investigator will be presented.

SECONDARY OUTCOMES:
Part 2: Percentage of Participants Who Experience an AE | Up to approximately 5 years
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The percentage of participants who experience AEs will be reported.
Part 2: Percentage of Participants Who Discontinue Study Treatment Due to an AE | Up to approximately 5 years
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The percentage of participants who discontinue study treatment due to an AE will be reported.
Part 1 and Part 2: Disease Control Rate (DCR) | Up to approximately 5 years
  DCR is defined, per RECIST 1.1, as the percentage of participants who have a CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions) or Stable Disease (SD). SD is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD: at least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm). Note: The appearance of one or more new lesions is also considered PD. The time from the first dose until the date of SD must be greater than or equal to 6 weeks. The DCR as assessed by the investigator will be presented.
Part 1 and Part 2: Time to Response (TTR) | Up to approximately 5 years
  For participants who demonstrate a confirmed CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1, TTR is defined as the time from the first dose to the first documented evidence of a CR or PR. The TTR as assessed by the investigator will be presented.
Part 1 and Part 2: Duration of Response (DOR) | Up to approximately 5 years
  For participants who demonstrate a confirmed CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1, DOR is defined as the time from first documented evidence of CR or PR until PD or death. PD is defined as at least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm. Note: The appearance of one or more new lesions is also considered PD. DOR as assessed by the investigator will be presented.
Part 1 and Part 2: Progression-free Survival (PFS) | Up to approximately 5 years
  PFS is defined as the time from randomization to the first documented PD or death due to any cause, whichever occurs first as assessed by RECIST 1.1. PD is defined as at least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm. Note: The appearance of one or more new lesions is also considered PD. PFS as assessed by the investigator will be presented.
Part 1 and Part 2: Overall Survival (OS) | Up to approximately 5 years
  OS is defined as time from first dose of study treatment to death due to any cause.
Part 2: AUC of total anti-HER3 antibody LC-MS in plasma | At designated timepoints (up to approximately 5 years)
  Blood samples will be collected at specified intervals for the determination of AUC.
Part 2: AUC of anti-HER3-ac-DXd in plasma | At designated timepoints (up to approximately 5 years)
  Blood samples will be collected at specified intervals for the determination of AUC.
Part 2: AUC of DXd in plasma | At designated timepoints (up to approximately 5 years)
  Blood samples will be collected at specified intervals for the determination of AUC.
Part 2: Cmax of anti-HER3 antibody LC-MS in plasma | At designated timepoints (up to approximately 5 years)
  Blood samples will be collected at specified intervals for the determination of Cmax.
Part 2: Cmax of anti-HER3-ac-DXd in plasma | At designated timepoints (up to approximately 5 years)
  Blood samples will be collected at specified intervals for the determination of Cmax.
Part 2: Cmax of DXd in plasma | At designated timepoints (up to approximately 5 years)
  Blood samples will be collected at specified intervals for the determination of Cmax.
Part 2: Ctrough of anti-HER3 antibody LC-MS in plasma | At designated timepoints (up to approximately 5 years)
  Blood samples will be collected at specified intervals for the determination of Ctrough.
Part 2: Ctrough of anti-HER3-ac-DXd in plasma | At designated timepoints (up to approximately 5 years)
  Blood samples will be collected at specified intervals for the determination of Ctrough.
Part 2: Ctrough of DXd in plasma | At designated timepoints (up to approximately 5 years)
  Blood samples will be collected at specified intervals for the determination of Ctrough.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (47):
- United States (13):
  - Children's Hospital Colorado-Center for Cancer and Blood Disorders ( Site 3016), Aurora, Colorado
  - Johns Hopkins All Children's Hospital ( Site 3025), St. Petersburg, Florida
  - University of Iowa Health Care Holden Comprehensive Cancer Center ( Site 3017), Iowa City, Iowa
  - Corewell Health ( Site 3001), Grand Rapids, Michigan
  - Children's Mercy Hospital ( Site 3024), Kansas City, Missouri
  - Rutgers Cancer Institute of New Jersey ( Site 3008), New Brunswick, New Jersey
  - New York Medical College ( Site 3023), Valhalla, New York
  - Sanford Fargo Medical Center-Roger Maris Cancer Center ( Site 3003), Fargo, North Dakota
  - Oregon Health and Science University ( Site 3004), Portland, Oregon
  - Children's Hospital of Philadelphia (CHOP) ( Site 3021), Philadelphia, Pennsylvania
  - Sanford Children's Hospital ( Site 3015), Sioux Falls, South Dakota
  - University of Texas-MD Anderson Cancer Center ( Site 3007), Houston, Texas
  - Intermountain - Primary Children's Hospital ( Site 3014), Salt Lake City, Utah
- Australia (2):
  - Sydney Children's Hospital-Kids Cancer Centre ( Site 3997), Sydney, New South Wales
  - Queensland Children's Hospital ( Site 3996), Brisbane, Queensland
- UZ Gent ( Site 3428), Ghent, Oost-Vlaanderen, Belgium
- Fundação Pio XII - Hospital de Câncer de Barretos ( Site 3264), Barretos, São Paulo, Brazil
- Colombia (3):
  - Hospital Pablo Tobon Uribe ( Site 3923), Medellín, Antioquia
  - Clinica de la Costa S.A.S. ( Site 3924), Barranquilla, Atlántico
  - IMAT S.A.S ( Site 3921), Montería, Departamento de Córdoba
- Czechia (2):
  - Detska nemocnice FN Brno ( Site 3388), Brno, Brno-mesto
  - Fakultni nemocnice v Motole-Klinika detske hematologie a onkologie ( Site 3387), Prague, Praha 5
- Rigshospitalet-Department of paediatrics and adolescent medicine, Section of Paed haem-onc ( Site 3467), Copenhagen, Capital Region, Denmark
- France (4):
  - Bordeaux University Hospital - Pellegrin ( Site 3105), Bordeaux, Aquitaine
  - Assistance Publique Hôpitaux de Marseille - Hôpital de la Timone ( Site 3102), Marseille, Bouches-du-Rhone
  - Centre Hospitalier Universitaire de Nantes - Hôpital Femme-Enfant-Adolescent Chu De Nantes ( Site 3104), Nantes, Loire-Atlantique
  - Centre Leon-Berard ( Site 3100), Lyon, Rhone
- Universitätsklinikum Münster - Albert Schweitzer Campus ( Site 3141), Münster, North Rhine-Westphalia, Germany
- Aghia Sophia Children's Hospital-First Department of Pediatrics, National and Kapodistrian Universi ( Site 3797), Athens, Attica, Greece
- Semmelweis University ( Site 3838), Budapest, Pest County, Hungary
- Israel (2):
  - Rambam Health Care Campus ( Site 3674), Haifa
  - Sheba Medical Center ( Site 3675), Ramat Gan
- Italy (3):
  - Fondazione IRCCS Istituto Nazionale dei Tumori ( Site 3552), Milan
  - Ospedale Pediatrico Bambino Gesù IRCCS ( Site 3553), Roma
  - Ospedale Infantile Regina Margherita ( Site 3551), Torino
- Prinses Maxima Centrum voor Kinderoncologie ( Site 3510), Utrecht, Netherlands
- Narodny ustav detskych chorob ( Site 3592), Bratislava, Bratislava Region, Slovakia
- South Korea (2):
  - Seoul National University Hospital-Pediatrics ( Site 3972), Seoul
  - Asan Medical Center-Pediatrics - Pedicatric Oncology ( Site 3973), Seoul
- Spain (3):
  - Hospital Sant Joan de Déu ( Site 3717), Esplugues de Llobregat, Barcelona
  - Hospital Universitari Vall d''Hebron ( Site 3716), Barcelona
  - Hospital Infantil Universitario Nino Jesus ( Site 3715), Madrid
- Sahlgrenska Universitetssjukhuset ( Site 3634), Gothenburg, Västra Götaland County, Sweden
- National Taiwan University Hospital ( Site 3983), Taiwan, Taipei, Taiwan
- Hacettepe Universitesi Tip Fakultesi Hastanesi ( Site 3961), Ankara, Turkey (Türkiye)
- United Kingdom (2):
  - Royal Victoria Infirmary ( Site 3348), Newcastle upon Tyne, England
  - University Hospital of Wales ( Site 3346), Cardiff

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com